CLINICAL TRIAL: NCT07395440
Title: A Prospective Observational Comparison of Quadratus Lumborum Block Techniques in Gynecologic Surgery
Brief Title: Comparison of Quadratus Lumborum Block Types in Open Gynecologic Surgery
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, KADİR TEOMAN, Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2025-068
Record Dates: First submitted 2025-04-19; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Pain Management; Gynecologic Surgical Procedures; Quadratus Lumborum Block
Keywords: quadratus lumborum block; open gynecological operations; acute pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to evaluate the effectiveness of Quadratus Lumborum Type 1 and Type 2 blocks on postoperative acute pain in gynecological operations performed with a Pfannenstiel incision.

DETAILED DESCRIPTION:
This prospective observational study was conducted to observe and analyze postoperative acute pain outcomes in patients undergoing open gynecologic surgery with a Pfannenstiel incision. The study included patients who received quadratus lumborum block (QLB) techniques as part of routine perioperative analgesic management.

Quadratus lumborum blocks were performed using ultrasound guidance according to standard clinical practice. The block was administered with the patient in the lateral position, and a high-frequency linear ultrasound transducer was used to identify the quadratus lumborum muscle and surrounding anatomical structures. For Quadratus Lumborum Type 1 (lateral) block, local anesthetic was injected at the anterolateral border of the quadratus lumborum muscle. For Quadratus Lumborum Type 2 (posterior) block, local anesthetic was deposited posterior to the quadratus lumborum muscle, within the thoracolumbar fascial plane.

The selection of Quadratus Lumborum Type 1 or Type 2 block was determined solely by the attending anesthesiologist based on routine clinical considerations, surgical characteristics, and patient-related factors. No intervention or regional analgesia technique was assigned by the investigators for the purpose of this study, and study participation did not influence anesthetic management. Participants would have received the same anesthetic and regional analgesia techniques in the same manner and intensity regardless of study enrollment.

Postoperative acute pain outcomes were prospectively collected and analyzed between predefined exposure groups according to the routinely applied quadratus lumborum block technique. The investigators did not modify clinical practice, dosing, timing, or performance of regional anesthesia. All anesthetic and analgesic interventions were provided as part of standard medical care.

This study was approved by the local ethics committee as an observational study and was conducted in accordance with institutional standards of care.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Female patients aged 18-80
* Cases undergoing open myomectomy and total abdominal hysterectomy

Exclusion Criteria:

* Those who do not want a block
* Patients who are allergic to local anesthetics
* Patients with coagulopathy
* Pregnancy
* Previous surgery in the area where the block will be applied

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who underwent open gynecological surgery
Study Population: female patients undergoing open gynecological surgery
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Reduction of opioid requirement in patients undergoing open myomectomy and total abdominal hysterectomy | from april to may
  It investigates the effectiveness of quadratus lumborum 1 block alone in acute pain, compared to quadratus lumborum 1 and 2 blocks applied together in patients undergoing open myomectomy and total abdominal hysterectomy.

SECONDARY OUTCOMES:
no need for additional analgesia | from 1 may to 15 may
  the first postoperative analgesic consumption in patients undergoing open myomectomy and total abdominal hysterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: KADİR T ETİKCAN, MEDİCAL DOCTOR, Principal Investigator — ANKARA ETLİK CİTY HOSPİTAL
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koksal E, Aygun H, Genc C, Kaya C, Dost B. Comparison of the analgesic effects of two quadratus lumborum blocks (QLBs), QLB type II vs QLB type III, in caesarean delivery: A randomised study. Int J Clin Pract. 2021 Oct;75(10):e14513. doi: 10.1111/ijcp.14513. Epub 2021 Jun 23. PMID 34117829
- [Result] Postoperative analgesic effects of the quadratus lumborum block III and transversalis fascia plane block in paediatric patients with developmental dysplasia of the hip undergoing open reduction surgeries: a double- blinded randomised controlled trial Congcong Huang,1,2 Xiaoguang Zhang,3 Chaoxuan Dong,4 Chunwei Lian Jun Li,2 Lingzhi Yu
- [Result] Bilgin S, Aygun H, Genc C, Dost B, Tulgar S, Kaya C, Sertoz N, Koksal E. Comparison of ultrasound-guided transversalis fascia plane block and anterior quadratus lumborum block in patients undergoing caesarean delivery: a randomized study. BMC Anesthesiol. 2023 Jul 21;23(1):246. doi: 10.1186/s12871-023-02206-w. PMID: 37480008; PMCID: PMC10362577.